CLINICAL TRIAL: NCT06784050
Title: Impact of Two Occlusal Schemes in Implant Retained Mandibular Overdenture on the Masticatory Efficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma ElSayed, assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00012891#133
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Edentulous Alveolar Ridge
Keywords: dental implant overdenture; occlusal scheme; masticatory efficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bilateral Balanced Occlusion Group (Active Comparator): This group received dentures designed with a bilateral balanced occlusion scheme. This occlusion scheme aims for simultaneous contact of teeth across the dental arch during jaw movements, purported to enhance stability and comfort.
  Interventions: Procedure: Bilateral Balanced Occlusion
- Monoplane Occlusion Group (Experimental): This group received dentures designed with a monoplane occlusion scheme. This scheme involves a flat occlusal plane without curvature, intended to reduce the complexity of denture fabrication and potentially improve masticatory efficiency by simplifying the occlusal contacts
  Interventions: Procedure: Monoplane Occlusion

INTERVENTIONS:
Procedure: Bilateral Balanced Occlusion — Dentures designed under this scheme feature a fully bilateral balanced articulation, ensuring bilateral, simultaneous contact of the anterior and posterior denture teeth in both centric and eccentric positions. This occlusal scheme is aimed at promoting stability and functionality of the dentures during various mandibular movements.
  Arms: Bilateral Balanced Occlusion Group
Procedure: Monoplane Occlusion — This scheme utilizes zero-degree teeth to create a flat occlusal plane, which is designed to simplify the occlusal contacts and minimize the transmission of lateral forces during mastication. The aim is to improve masticatory efficiency by reducing the complexity of tooth contact
  Arms: Monoplane Occlusion Group

SUMMARY:
Purpose: To assess the effect of two different occlusal schemes, bilateral balance and monoplane on the masticatory efficiency in mandibular implant retained overdenture with ball and socket attachment. Methodology: Twelve male completely edentulous patients were recruited for this clinical study. Each patient received two implants after that. Patients were divided randomly into two equal groups according to occlusal schemes which involved bilateral balanced occlusion and mono plane occlusion. each. Group 1 received a bilateral balanced occlusion scheme denture; Group 2 received monoplane occlusal scheme denture. Masticatory efficiencies were evaluated by assessing chewing time and number of chewing strokes with different types of foods. The data were collected, tabulated and statistically analyzed. Results: using dentures with bilateral balanced occlusion showed lower masticatory efficiency than the denture with monoplane occlusion with no significant difference when using soft food during the first month, while after 3 months there were significant differences between the two groups. Conclusion: The two-implant retained mandibular overdenture with monoplane occlusion showed relatively improved masticatory efficiency than with bilateral balanced occlusion.

DETAILED DESCRIPTION:
Dental research has shown that implant-retained overdentures markedly improve the quality of life for edentulous patients [1]. Research has shown that two dental implants are sufficient to support a mandibular overdenture [2]. Considering the increasingly old age and systemic health complications of these patients, it is imperative that dental implant treatment include minimum intervention for both surgical and prosthetic maintenance after the delivery of the final prosthesis. This requires reducing the transmission of stress to the dental implants via the overdenture and its framework, hence assuring fewer maintenance procedures [3].

The attachment systems used in implant-retained overdentures may be categorized according to the splinting of the implants. The connection between the prosthesis and the implant is made using bar structures when dental implants are splinted. If the dental implants are not splinted, each implant is independently affixed to the prosthetic structure using technologies such as Locator, ERA, ball, O-ring, and different magnetic systems.[1] The choice of attachment type is influenced by the location of the dental implant, the required degree of retention, the morphology of the edentulous jaw, and the patient's motor dexterity. The preferred attachment types for overdentures are the Locator and ball systems due to their ease of application, minimal technical requirements, and lower costs compared to bar or magnet systems. There is ongoing research and development to improve attachment systems in dental implantology. [2] The occlusal scheme for overdentures affects the pattern of occlusal contact between opposing teeth during centric relation and mandibular functional movements. Consequently, the quantity and intensity of these contacts are crucial in determining the overall efficacy and comfort of the prosthesis. [3] The occlusal scheme known as fully bilateral balanced articulation is designed to ensure bilateral, simultaneous contact of the anterior and posterior denture teeth in both centric and eccentric positions. This scheme aims to achieve a cross-arch balanced articulation, promoting stability and functionality for the dentures during various mandibular movements.[4] On the other hand, the monoplane concept, first proposed by De Van in 1954, utilizes zero-degree teeth and creates a perfectly flat occlusal plane that is parallel to and evenly divides the upper and lower residual ridges. The occlusal plane is positioned at the junction of the upper and middle third of the retromolar pad. This approach eliminates inclined planes both in the tooth form and the occlusal plane, ensuring that no lateral components are generated with vertical chewing forces.[5] Masticatory performance refers to the ability to triturate food under controlled testing settings. [9] These food crushing tests are designed to evaluate the fragmentation of test specimens into smaller fragments. The test specimens may consist of natural food products, such as carrots or nuts, or synthetic materials like silicone-based Optosil cubes or fuchsin beads .[6] Masticatory efficiency is the primary indicator of mastication function and reflects the functional potential of the dental system, including dentures. Assessment the masticatory efficiency is vital for a comprehensive evaluation of treatment outcomes involving implant-retained overdentures.[7] Electromyographic devices are research equipment for evaluating the electrical activity of the muscles. The behavior of masticatory muscles and information as to the functional state of the stomatognathic neuromuscular system can be obtained by electromyography. It is a practical and efficient method for the study of muscle function and activity, thus serving as a valuable tool in dental research

ELIGIBILITY:
Inclusion Criteria:

Male patients Completely edentulous Ages range from 55-60 years Residual alveolar ridges of maxilla and mandible covered by healthy, firm, compressible mucosa Free from any temporomandibular joint disorders Have Angle's class I jaw relation Edentulous mandible for at least 6 months No bone augmentation requirement Good oral hygiene

Exclusion Criteria:

Presence of any systemic conditions that could compromise implant surgery History of chemotherapy or radiotherapy to the head and neck region History of taking bisphosphonates Heavy smoker status

Ages: 55 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-09-22 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Masticatory Efficiency Using Soft Food | Assessments were made at three points, baseline, after one month and three months from the start of using the overdentures.
  The masticatory efficiency was assessed by measuring the number of chewing strokes and the time taken to achieve the first swallow and complete mouth clearance while chewing standardized pieces of soft food.
Masticatory Efficiency Using Hard Food | Assessments were made at three points, baseline, after one month and three months from the start of using the overdentures.
  Similar to the soft food assessment, the efficiency for chewing hard food was evaluated by counting the number of chewing strokes and timing the duration until the first swallow and until the mouth was cleared of food.

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient clinic of the Prosthodontic Department, Faculty of Oral and Dental Medicine, Ahram Canadian University., Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided